CLINICAL TRIAL: NCT05729815
Title: Effects of Three Body-oriented Intervention Programs on Preschoolers' Social-emotional Competence
Brief Title: Body-oriented Interventions on Preschoolers' Social-emotional Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Andreia Dias Rodrigues, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOICHI28122022
Record Dates: First submitted 2022-12-28; First posted 2023-02-15 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Social-emotional Competence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Relaxation group (Experimental): Relaxation program sessions had 3 phases: initial dialogue (2 min); a main section (25 min); final ritual (3 min). During the main section, participants listened and observed the therapist, who described and demonstrated all the exercises of the session, which were focused on Jacques Choque Method (Choque, 1994).
  Interventions: Other: Relaxation
- Loose parts play group (Experimental): Loose Parts Play program sessions had 3 phases: initial dialogue (2 min); main section (25 min); final ritual (3 min). During the main section, participants were allowed to play freely with any materials (loose parts) available in the playground.
  Interventions: Other: Loose parts play
- Combined group (Experimental): In the combined program, the sessions had 4 phases: initial dialogue (3 min); loose parts play moment (20 min); relaxation exercises moment (5 min); final ritual (2 min).
  Interventions: Other: Combined
- Control group (No Intervention): No intervention. Maintained their usual routines.

INTERVENTIONS:
Other: Relaxation — Sessions focused on relaxations activities (Jacques Choque Method).
  Arms: Relaxation group
Other: Loose parts play — Loose parts play-based sessions, with open-ended materials.
  Arms: Loose parts play group
Other: Combined — Sessions focused on loose parts play and relaxation activities.
  Arms: Combined group

SUMMARY:
Experimental study with 4 groups (3 experimental and 1 control). Examine the effects of 3 body-oriented intervention programs on preschoolers' social-emotional competence.

Intervention programs focused on relaxation, loose parts play and combined loose parts play and relaxation, for 12 weeks with 2 30-min sessions per week.

DETAILED DESCRIPTION:
To examine the chronic effects of the intervention programs, instruments were collected at baseline (pretest) and at the end of the 12-week period (post-test). To measure the acute effects, salivary cortisol was measured at the beginning and end of the 1st and the 24th sessions.

ELIGIBILITY:
Inclusion Criteria:

* participants' age between 3 and 6 years
* do not have participated in a similar intervention program within the last 6 months
* do not have a physical condition that can affect the participation in the program.

Exclusion Criteria:

* participants' age less than 3 and under 6 years
* have participated in a similar intervention program within the last 6 months
* have a physical condition that can affect the participation in the program.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Change in Emotion discrimination | 1 and 12 weeks
  Emotion discrimination was measured through the Emotion-discrimination Task. This measurement consists in two performance tasks of increasing difficulty. In the task 1 (neutral condition) children were tested on their ability to discriminate between cars and flowers, and faces with hats versus faces with glasses. This neutral condition is not scored, since is used to check if children understood how to sort different cards. In task 2, children had a sheet in front of them with a sample drawing of one category in the top left corner (e.g. an angry face) and a drawing of the other category in the top right corner (e.g. a sad face). Then, children have six cards (with the same emotion) and one by one they have to place each card in the correct category after a demonstration. The cards that were placed correctly were counted with 1 point, with a maximum of 3 points.
Change in Emotion identification | 1 and 12 weeks
  Emotion identification was measured through the Emotion-identification Task. The task consists of eight drawings of facial emotion expressions, two for each emotion (happiness, sadness, fear, and anger). Then the researcher show two sheets with four drawings of facial emotion expressions on each sheet and ask to the children: "Who looks happy?", and children have to point to the drawing with the correct facial expression. Next, the researcher ask if "Is there anybody else who looks happy?". This procedure is repeated for anger, sadness, and fear. The number of emotions correctly identified was recorded, with a maximum score of 2 per emotion.
Change in Emotion recognition | 1 and 12 weeks
  Emotion recognition was measured thought the subscale Others' Emotion Recognition (6 items) of the Portuguese version of the Emotion Expression Questionnaire. This Subscale indicates the extent to which the child can recognise the parents' and others' emotions. Parents can rate to what degree each item is true on a 5-point scale (0=(almost) never, 1=rarely, 2=sometimes, 3=often, 4=(almost) always).
Change in Positive and negative emotion expression | 1 and 12 weeks
  Positive emotion expression, and negative emotion expression was measured through the Negative Emotion Expression subscale (8 items) and Positive Emotion Expression subscale (6 items) from the EEQ. Parents scored on a 5-point scale (0=(almost) never, 1=rarely, 2=sometimes, 3=often, 4=(almost) always), the frequency, intensity, and duration of child's expressions of negative emotions (e.g., anger, sadness), and positive emotions (e.g., happiness, joy). The extent to which the child can calm down from the emotional episode was also measured (1=easy; 3= difficult).
Change in Self-regulation | 1 and 12 weeks
  Self-regulation was measured through the Portuguese version of Head-Toes-Knees-Shoulders Task (HTKS). Using no materials, the HTKS has three sections with up to four paired behavioral rules: "touch your head" and "touch your toes"; "touch your shoulders" and "touch your knees". Child first respond naturally, but then had to perform the opposite of a dominant response (e.g., touch your head when the interviewer says "touch your toes"). This task includes three phases (each with 10 trials), and for each trial, the child received a score of 0 (incorrect), 1 (self-correct), or 2 (correct).
Change in Stress regulation | 2 days
  Stress regulation was measured through cortisol levels (mcg/dL) was quantified in saliva samples collected at the same time and in the same place where the interventions occurred, before and after the 1st and 24th sessions. Samples were collected directly from each child's mouth, without stimulation, by passive droll during 5 minutes to a polyethylene tube.
Change in Social competence | 1 and 12 weeks
  Social competence was obtained through the prosocial behaviors scale (5 items), and positive items from the peer problems scale (2 items) of the Portuguese version of Strengths and Difficulties Questionnaire (SDQ). Rated on a 3-point scale (0 = not true, 1 = somewhat true, and 2 = certainly true) the degree to which each item represented child's behavior in the last 3 months.
Change in Externalizing problems | 1 and 12 weeks
  Externalizing problems was obtained also through the behavior problems scale (5 items), and hyperactivity scale (5 items) of the Strengths and Difficulties Questionnaire (SDQ). Rated on a 3-point scale (0 = not true, 1 = somewhat true, and 2 = certainly true) the degree to which each item represented child's behavior in the last 3 months.
Change in Conflicts resolution | 1 and 12 weeks
  Conflicts resolution was measured through the conflict resolution strategies subscale (6 items) of the Portuguese version of Social Strategies Rating Scale (SSRS). Administered to teachers, which rated on a 5-point scale (1=never, 3=half of the time, 5=almost always) how often the child uses the social strategies during interactions with peers on preschool context.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia D Rodrigues, Principal Investigator — PhD student
Locations (1):
- Andreia Dias Rodrigues, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05729815/ICF_000.pdf